CLINICAL TRIAL: NCT05600621
Title: Suubi+Adherence4Youth: Optimizing the Suubi Intervention for Adherence to HIV Treatment for Youth Living With HIV in Uganda
Brief Title: Suubi+Adherence4Youth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Fred Ssewamala, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01MH131507 (NIH)
Record Dates: First submitted 2022-10-05; First posted 2022-10-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: HIV
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The factorial experiment is guided by the Multiphase Optimization Strategy (MOST).
  The 4 intervention components are:
  Component 1. Financial Literacy Training (FLT); Component 2. Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs); Component 3. A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon); Component 4. Engagement with HIV treatment-experienced role models who share their lived experiences of HIV.
  Clinics will be randomized to provide one of the 16 conditions, with 12 ALHIV (aged 11-17 years) enrolled per clinic, yielding main effects and interaction effects for the 4 components on sustained viral suppression.
Who Masked: Participant
Masking Description: Participants will be blinded to the experimental condition that the participant was assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1: Components 1, 2,3 and 4 (Experimental): Participants will be assigned to receive all of the four intervention programs:
  1. Financial Literacy Training (FLT) Workshops
  2. Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs)
  3. A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon)
  4. Engagement with HIV treatment-experienced role models who share lived experiences of HIV.
  Interventions: Behavioral: Financial Literacy Training (FLT) Workshops; Behavioral: Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs); Behavioral: A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon).; Behavioral: Engagement with HIV treatment-experienced role models who share lived experiences of HIV
- Condition 2: Components 1, 2 and 3 (Experimental): 1. Financial Literacy Training (FLT) Workshops
  2. Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs)
  3. A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon)
  Interventions: Behavioral: Financial Literacy Training (FLT) Workshops; Behavioral: Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs); Behavioral: A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon).
- Condition 3: Components 1, 2 and 4 (Experimental): 1. Financial Literacy Training (FLT) Workshops
  2. Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs)
  4.Engagement with HIV treatment-experienced role models who share lived experiences of HIV.
  Interventions: Behavioral: Financial Literacy Training (FLT) Workshops; Behavioral: Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs); Behavioral: Engagement with HIV treatment-experienced role models who share lived experiences of HIV
- Condition 4: Components 1 and 2 (Experimental): 1. Financial Literacy Training (FLT) Workshops
  2. Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs)
  Interventions: Behavioral: Financial Literacy Training (FLT) Workshops; Behavioral: Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs)
- Condition 5: Components 1,3 and 4 (Experimental): 1.Financial Literacy Training (FLT) Workshops
  3.A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon)
  4.Engagement with HIV treatment-experienced role models who share lived experiences of HIV.
  Interventions: Behavioral: Financial Literacy Training (FLT) Workshops; Behavioral: A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon).; Behavioral: Engagement with HIV treatment-experienced role models who share lived experiences of HIV
- Condition 6: Components 1 and 3 (Experimental): 1.Financial Literacy Training (FLT) Workshops
  3.A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon)
  Interventions: Behavioral: Financial Literacy Training (FLT) Workshops; Behavioral: A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon).
- Condition 7: Components 1 and 4 (Experimental): 1.Financial Literacy Training (FLT) Workshops
  4.Engagement with HIV treatment-experienced role models who share lived experiences of HIV.
  Interventions: Behavioral: Financial Literacy Training (FLT) Workshops; Behavioral: Engagement with HIV treatment-experienced role models who share lived experiences of HIV
- Condition 8: Components 1 (Experimental): 1.Financial Literacy Training (FLT) Workshops
  Interventions: Behavioral: Financial Literacy Training (FLT) Workshops
- Condition 9: Components 2,3 and 4 (Experimental): 2.Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs)
  3.A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon)
  4.Engagement with HIV treatment-experienced role models who share lived experiences of HIV.
  Interventions: Behavioral: Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs); Behavioral: A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon).; Behavioral: Engagement with HIV treatment-experienced role models who share lived experiences of HIV
- Condition 10: Components 2 and 3 (Experimental): 2.Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs)
  3.A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon)
  Interventions: Behavioral: Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs); Behavioral: A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon).
- Condition 11: Components 2 and 4 (Experimental): 2.Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs)
  4.Engagement with HIV treatment-experienced role models who share lived experiences of HIV.
  Interventions: Behavioral: Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs); Behavioral: Engagement with HIV treatment-experienced role models who share lived experiences of HIV
- Condition 12: Components 2 (Experimental): 2.Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs)
  Interventions: Behavioral: Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs)
- Condition 13: Components 3 and 4 (Experimental): 3.A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon)
  4.Engagement with HIV treatment-experienced role models who share lived experiences of HIV.
  Interventions: Behavioral: A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon).; Behavioral: Engagement with HIV treatment-experienced role models who share lived experiences of HIV
- Condition 14: Components 3 (Experimental): 3.A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon)
  Interventions: Behavioral: A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon).
- Condition 15: Components 4 (Experimental): 4.Engagement with HIV treatment-experienced role models who share lived experiences of HIV.
  Interventions: Behavioral: Engagement with HIV treatment-experienced role models who share lived experiences of HIV
- Condition 16: No Components (Experimental): Participants not assigned to any of the 4 components
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Financial Literacy Training (FLT) Workshops — Participants will be assigned to receive FLT workshops which are implemented by community-level agencies in collaboration with the financial institutions. FLT comprises six workshops delivered over 6 weeks. Topics include: a) an introduction to the notion of asset-building; b) coverage of asset-building strategies in detail, e.g., saving; c) coverage of specific topics related to saving, e.g., the importance of saving and how to save, d) an introduction of banking services to participants and e) coverage of basics of borrowing and debt management. Participants from the same location, in this case, clinics are assigned to the same group. Workshops occur on weekends to accommodate participants week-day schedules, including school and/or gardening.
  Arms: Condition 1: Components 1, 2,3 and 4; Condition 2: Components 1, 2 and 3; Condition 3: Components 1, 2 and 4; Condition 4: Components 1 and 2; Condition 5: Components 1,3 and 4; Condition 6: Components 1 and 3; Condition 7: Components 1 and 4; Condition 8: Components 1
Behavioral: Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs) — ALHIV will receive a YSA with a 1:1 matched savings program at a financial institution accredited by the Bank of Uganda. Each YDA will be opened in the name of the adolescent, with their primary caregiver as a co-signer, until the adolescent turns 18 years. The account will then be matched with money from the program on 1:1 rate.
  As part of YSA, ALHIV are also trained on investing in income-generating activities (IGA) and are normally allowed to use up to 30% of their matched savings to invest in an IGA to benefit their family. The IGA portion helps promote economic stability for families and enable the ALHIV to afford medical expenses.
  Arms: Condition 10: Components 2 and 3; Condition 11: Components 2 and 4; Condition 12: Components 2; Condition 1: Components 1, 2,3 and 4; Condition 2: Components 1, 2 and 3; Condition 3: Components 1, 2 and 4; Condition 4: Components 1 and 2; Condition 9: Components 2,3 and 4
Behavioral: A manualized visual-based intervention for ART adherence and stigma reduction using multiple family group approach (Suubi Cartoon). — Participants assigned to this component will participate together with her/his caregiving family, in attending sixteen 60 minute sessions hosted within the community over 16 weeks. Each session involves 6-10 families. Participants will learn from the Suubi Cartoon curriculum about their HIV diagnosis and treatment needs, while coping with family loss, stigma, peer relationships, identity, and family functioning.
  Arms: Condition 10: Components 2 and 3; Condition 13: Components 3 and 4; Condition 14: Components 3; Condition 1: Components 1, 2,3 and 4; Condition 2: Components 1, 2 and 3; Condition 5: Components 1,3 and 4; Condition 6: Components 1 and 3; Condition 9: Components 2,3 and 4
Behavioral: Engagement with HIV treatment-experienced role models who share lived experiences of HIV — Participants will be assigned to small groups with an average of 3-4 peers from the same health clinic, and each ALHIV stays in the same group -- for 9 sessions - with the same role model. This is intended to build trust and rapport not only between the role model and mentee, but also between all group members. The 9 sessions, to be conducted over a 6-month period, include activities, videos, scenarios, and role-playing to facilitate discussion and learning. This is intended to promote their self-esteem, improve their HIV care engagement, reduce stigma and stress, encourage hopefulness, build stronger communication skills with their caregivers and/or family members, enhance safe sexual decision-making, and decrease sexual risk-taking behavior.
  Arms: Condition 11: Components 2 and 4; Condition 13: Components 3 and 4; Condition 15: Components 4; Condition 1: Components 1, 2,3 and 4; Condition 3: Components 1, 2 and 4; Condition 5: Components 1,3 and 4; Condition 7: Components 1 and 4; Condition 9: Components 2,3 and 4
Other: Standard of Care (SOC) — SOC consisting of pediatric ART initiation and monitoring outlined by Uganda's Ministry of Health.
  Arms: Condition 16: No Components

SUMMARY:
The study will test four economic empowerment intervention components to identify the combination that best enhance viral suppression.

The study design is a 2-to-the 4 factorial experiment. The 2 represents the level of each component:0 (receive) or (don't receive) four components: 1) Financial Literacy Training (FLT); 2) Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs); 3) A manualized intervention for ART adherence and stigma reduction (Suubi Cartoon); and 4) Engagement with HIV treatment-experienced role models who share their lived experiences of HIV. Guided by the MOST framework, the study will test each of the four components' performance and their combinations on the primary outcome, viral suppression. Resulting in 16 unique conditions representing all possible combinations of the 4 components. The study will randomize at the level of health clinics (N=48). Clinics will be randomized to provide one of the 16 conditions, with 12 ALHIV (aged 11-17 years) enrolled per clinic, yielding main effects and interaction effects for the 4 components on sustained viral suppression. Sustained viral suppression is defined as an undetectable viral load on all 12-, 24- and 36-month follow-up assessments.

DETAILED DESCRIPTION:
The number of adolescents living with HIV (ALHIV) in Uganda is over 170,000 and growing. Ugandan ALHIV are a priority due to social and structural inequities that make them highly vulnerable to HIV infection and sub-optimal access and adherence to antiretroviral therapy (ART). Less than 50% of ALHIV in Uganda are ART-adherent leading to low rates of viral suppression and high rates of attrition from HIV care. In response to the call for expanding differentiated care approaches for ALHIV and new forms of combination HIV interventions, we seek to intervene on social and structural inequities as economic and psychosocial hardships exacerbate the risk for viral load non-suppression. Addressing these hardships can improve the livelihoods of ALHIV and give them the knowledge and resources to sustainably manage HIV.

With 15+ years of intervention research combining 1) economic empowerment (EE) and 2) psychosocial components for HIV prevention, care and support for adolescents in SSA, we have demonstrated the effectiveness of Suubi (Hope), our multi-component combination intervention tested in four RCTs in Uganda (R01HD070727, R01HD074949, R34MH081763, R01MH113486) and one foundation-funded study in Kenya. With EE components to address economic hardships and psychosocial components to address ART non-adherence and HIV stigma, we have improved viral suppression and psychosocial and mental health functioning. Suubi is evidence-based and theory-informed and has four components: 1) Financial Literacy Training (FLT); 2) Incentivized Matched Youth Savings Accounts (YSA) with income-generating activities (IGAs); 3) A manualized intervention for ART adherence and stigma reduction (Suubi Cartoon); and 4) Engagement with HIV treatment-experienced role models who share their lived experiences of HIV. Suubi has shown robust effects on viral suppression and ART adherence, mental health, psychosocial outcomes, and family financial stability and cohesion. However, it is unknown if each component in Suubi had a positive effect, how the components interacted, or if fewer components could have produced equivalent effects. Given our successes and infrastructure, we are well-positioned to unpack and optimize Suubi to identify the most impactful and sustainable components for scale up across Uganda.

The study will use a factorial experiment to unpack, test, and optimize the Suubi intervention to enhance scale up in health systems using the multi-phase optimization strategy (MOST), an engineering-inspired intervention framework. Guided by the MOST framework, the study will test each of the four components' performance and their combinations in a fully powered efficient factorial experiment on the primary outcome, viral suppression. Then a pre-specified optimization objective will be set to create the new "optimized" intervention. We define our "optimization objective" as the most cost-effective components that addresses three real-world constraints (i.e., challenges to implementation): 1) efficiency (do the components work within our existing health systems?), 2) affordability (do observed effect sizes justify costs and labor?), and 3) scalability (do components perform exactly as they would at scale?). The study will evaluate various component combination effect sizes and balance them against real-world constraints and costing data to empirically arrive at optimization. Our goal is to build Suubi 2.0 (hereafter, Suubi+Adherence4Youth), a combination of components for viral suppression that meets standards for being efficient, affordable, and working at scale.

The study will be guided by the following specific aims:

Aim 1. Conduct a factorial experiment (optimization trial) to test the main effects of each of the four Suubi intervention components and combinations of components (interactions) on viral suppression (primary outcome);

Aim 2. Test mediators and explore moderators that explain and modify the relationship between each of the four Suubi intervention components and viral suppression;

Aim 3. Compare the cost and cost-effectiveness of each of the four Suubi intervention components and every combination of components.

ELIGIBILITY:
Inclusion Criteria:

Adolescent:

* living with HIV (confirmed by medical report and aware of status)
* living within a family
* being 11-17 years of age (at enrollment)
* prescribed ART
* enrolled in ART care at one of the 48 health clinics in the study districts.

Health clinics would be eligible if they:

* have existing procedures tailored to adolescent adherence (including adolescent-specific clinic days and peer counselling)
* Accredited by the Uganda Ministry of Health as a provider of ART within the study districts.

Exclusion Criteria:

* Includes an inability to understand study procedures and participant rights as assessed during informed consent/assent process with the adolescent or parent.
* If the adolescent or adult caregiver presents with emergency needs (e.g., hospitalization), needed care will be secured, rather than study participation

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 576 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Achievement of Viral Suppression | Baseline 12, 24 and 36 month follow-up
  Change in viral suppression will be assessed using viral load (VL) data collected from health clinic records. VL will be dichotomized between undetectable /suppression (VL< 40 copies/ml) and detectable/failed viral suppression (VL > =40 copies/ml) levels at each assessment time.
Cost-Effectiveness Analyses | Baseline 12, 24 and 36 month follow-up
  Cost-effectiveness analyses measuring the cost of achieving an agreed upon benefit, such as cost of staff time, supplies, overhead of IDA's, as measured by admin review and project records.

SECONDARY OUTCOMES:
Financial Literacy | Baseline 12, 24 and 36 month follow-up
  Change in Financial Literacy knowledge will be measured using the Financial Literacy Knowledge item, with higher scores indicating higher financial literacy.
Financial management skills | Baseline 12, 24 and 36 month follow-up
  Change in financial management skills will be measured using the Attitudes about Saving Scale, with higher scores indicating greater financial management skills.
Engagement with financial institutions | Baseline 12, 24 and 36 month follow-up
  Change in engagement with financial institutions will be measured using the frequency of deposits and withdrawals by data from bank statements.
Change in confidence to save | Baseline 12, 24 and 36 month follow-up
  Change in confidence to save will be measured using the Financial Literacy Knowledge item, with higher scores indicating higher confidence to save.
Change in motivation to save | Baseline 12, 24 and 36 month follow-up
  Motivation to save will be measured using the Financial Literacy Knowledge item, with higher scores indicating higher motivation to save.
Change in savings amount and Investment in IGA | Baseline 12, 24 and 36 month follow-up
  Change in savings amount and investment measured by data from bank statements

OTHER OUTCOMES:
Change in ART knowledge and ART adherence | Baseline 12, 24 and 36 month follow-up
  Change in adolescent Self reported medication adherence. This will be measured using the Adherence and retention in care questionnaire focusing on the pharmacy refills, pill counts and missed appointments at each assessment time.
Reductions in internalized stigma | Baseline 12, 24 and 36 month follow-up
  Reductions in internalized stigma will be measured using the Social Impact Scale on a range of 24 - 96, with higher scores indicating higher levels of internalized stigma.
Sexual negotiation and communication skills | Baseline 12, 24 and 36 month follow-up
  Ability to negotiate safe sex practices measured using the Sexual Communication Scale. Responses are summed and scored on a range of 20 - 100, with higher scores representing greater levels of communication.
Change in mental health-hopelessness symptoms | Baseline 12, 24 and 36 month follow-up
  Hopelessness will be measured using the Beck Hopelessness Scale. The study will assess the mean scores over time. The total score range is between 0 - 20, with a higher score indicating higher levels of child hopelessness.
Change in depressive symptoms | Baseline 12, 24 and 36 month follow-up
  Depression will be measured using the Center for Epidemiological Studies-Depression Scale (CES-D). The total score range is between 0 - 60, with higher scores indicating the presence of more symptomatology.
Change in HIV Stigma | Baseline 12, 24 and 36 month follow-up
  Change in HIV stigma will be measured using the Negative Self-image sub-scale of HIV Stigma Scale. The total score range is between 40 - 160 with higher scores indicating higher levels of perceived HIV-associated stigma.
Positive HIV Identity | Baseline 12, 24 and 36 month follow-up
  HIV Positive Identity Scale
Problem solving of HIV care logistics | Baseline 12, 24 and 36 month follow-up
  Self-reported questionnaires
Self-esteem | Baseline 12, 24 and 36 month follow-up
  Self esteem will be measured using Rosenberg Self-Esteem Scale. The study will assess the mean scores over time. The total score range between10 - 40, with a higher score indicating high levels of child self esteem.
Social support | Baseline 12, 24 and 36 month follow-up
  Change in social support will be measured by Social Support Behavior Scale.
Engagement and retention of HIV care metrics | Baseline 12, 24 and 36 month follow-up
  The degree to which a patient feels engaged/disengaged from HIV care will be measured using the HIV Index of Engagement on a range of 10 - 50, with higher scores indicating better engagement.

CONTACTS AND LOCATIONS:
Locations (1):
- International Center for Child Health and Development, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Once all of the data has been de-identified, cleaned, and validated, and main findings have been published, the Investigators expect to share data with the scientific community. The research team will make datasets available to any individual who makes a direct request to the PI and indicates the data will be used for the purposes of research (per Code of Federal Regulations Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge."). In sharing participant data, the team will follow Washington University in St. Louis' Office of Sponsored Projects' data sharing agreement.
Supporting Information: Study Protocol, Analytic Code

REFERENCES:
- [Derived] Ssewamala FM, Sauceda JA, Brathwaite R, Neilands TB, Nabunya P, Brown D, Sensoy Bahar O, Namuwonge F, Nakasujja N, Mugarura A, Mwebembezi A, Nartey P, Mukasa B, Gwadz M. Suubi + Adherence4Youth: a study protocol to optimize the Suubi Intervention for Adherence to HIV treatment for youth living with HIV in Uganda. BMC Public Health. 2023 Apr 20;23(1):717. doi: 10.1186/s12889-023-15564-4. PMID 37081534